CLINICAL TRIAL: NCT05404620
Title: Comparative Effects of Schroth Method and Proprioceptive Neuromuscular Facilitation Technique on Pain, Mobility and Quality of Life in Patients With Idiopathic Scoliosis
Brief Title: Effects of Schroth Method and Proprioceptive Neuromuscular Facilitation Technique in Patients With Idiopathic Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0121
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Idiopathic Scoliosis
Keywords: idiopathic scoliosis; schroth method; proprioceptive neuromuscular facilitation techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth exercises (Experimental): Mobilization in the spine between ribs will be performed to increase the mobility of joints. To strengthen the muscles such as erector spinae, iliopsoas, and the quadratus lumborum, muscle activation will be done. Then the four exercises of the Schroth method which are the "50 x Swiss ball" exercise, Prone exercise, Sail exercise, and the Muscle-cylinder exercise will be performed. This will be followed by hot pack and static stretching of muscles.
  Interventions: Other: Schroth exercises
- PNF technique (Experimental): This technique involves the specific program and pattern of PNF that are deep breathing, pelvic posterior tilting, DI flexion & Extension of UL and D2 flexion, and extension of LL. + Hot pack + static stretching of the involved muscles.
  Interventions: Other: PNF technique

INTERVENTIONS:
Other: Schroth exercises — 9 participants will perform Schroth exercises with 2 mint rest between each exercise. + Hot pack (10 mint) +static stretching of the involved muscles with 10 to 30-sec hold and 2 to 4 repetitions as a standard treatment. A total of 45 min sessions three times a week on alternate days for three weeks will be provided.
  Arms: Schroth exercises
Other: PNF technique — 9 participants will perform PNF techniques followed by a hot pack for 10 minutes and static stretching of the involved muscles with 10 to 30-sec hold and 2 to 4 repetitions as a standard treatment. A total of 45 min sessions three times a week on alternate days for three weeks will be given.
  Arms: PNF technique

SUMMARY:
The aim of this study is to compare the effects of schroth method and proprioceptive neuromuscular facilitation techniques on pain, mobility, and quality of life in patients with idiopathic scoliosis.

DETAILED DESCRIPTION:
Scoliosis is a three-dimensional deformity that causes the spine to curve sideways. The most common type of scoliosis is "idiopathic," which means the exact cause is unknown. It accounts for approximately 85% of cases. The prevalence rate of 2-5% with a Cobb angle greater than 10 degrees. All previous studies in which schroth method with other different techniques has been performed have shown greater improvement in the management of scoliosis. However, there is no clinical significance work on the Comparative effect of the schroth method and PNF. Previous literature showed no significant improvement in mobility and quality of life. This study aims to find evidence of clinical significance work on effects of Schroth method and proprioceptive neuromuscular facilitation technique on pain, mobility, and quality of life in patients with idiopathic scoliosis in both gender

ELIGIBILITY:
Inclusion Criteria:

* Participants with Lenke curve type 1 scoliosis and other types of scoliotic curve magnitude will be included.
* Cobb angle 10-30

Exclusion Criteria:

* Participants with any surgical and traumatic history of spine
* Participants prescribed with brace treatment
* Subjects with Non-idiopathic scoliosis
* Subjects with any systematic disease e.g. (cardiovascular, vestibular, rheumatological, neuromuscular and pulmonary disease)

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
NPRS for pain | 3rd week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Goniometer for range of motion | 3rd week
  It will be used to measure flexion, extension, and lateral flexion of the spine.
SRS-22 questionnaire for quality of life | 3rd week
  It includes five domains: self-image, function, pain, mental health (five questions each), and satisfaction with treatment (two questions) to assess the quality of life with scoliosis.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- GOVT EYE-CUM general hospital (THQ), Gojra, Gojra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- [Background] Lee HJ, Seong HD, Bae YH, Jang HY, Chae SH, Kim KH, Lee SM. Effect of the Schroth method of emphasis of active holding on Cobb's angle in patients with scoliosis: a case report. J Phys Ther Sci. 2016 Oct;28(10):2975-2978. doi: 10.1589/jpts.28.2975. Epub 2016 Oct 28. PMID 27821972
- [Background] Stepien A, Fabian K, Graff K, Podgurniak M, Wit A. An immediate effect of PNF specific mobilization on the angle of trunk rotation and the Trunk-Pelvis-Hip Angle range of motion in adolescent girls with double idiopathic scoliosis-a pilot study. Scoliosis Spinal Disord. 2017 Sep 6;12:29. doi: 10.1186/s13013-017-0132-0. eCollection 2017. PMID 28905003
- [Background] BECKERS DB. PNF in practice: an illustrated guide: SPRINGER-VERLAG BERLIN AN; 2020.
- [Background] Mohamed RA, Yousef AM. Impact of Schroth three-dimensional vs. proprioceptive neuromuscular facilitation techniques in adolescent idiopathic scoliosis: a randomized controlled study. Eur Rev Med Pharmacol Sci. 2021 Dec;25(24):7717-7725. doi: 10.26355/eurrev_202112_27618. PMID 34982433
- [Background] Kocaman H, Bek N, Kaya MH, Buyukturan B, Yetis M, Buyukturan O. The effectiveness of two different exercise approaches in adolescent idiopathic scoliosis: A single-blind, randomized-controlled trial. PLoS One. 2021 Apr 15;16(4):e0249492. doi: 10.1371/journal.pone.0249492. eCollection 2021. PMID 33857180
- [Background] Burger M, Coetzee W, du Plessis LZ, Geldenhuys L, Joubert F, Myburgh E, van Rooyen C, Vermeulen N. The effectiveness of Schroth exercises in adolescents with idiopathic scoliosis: A systematic review and meta-analysis. S Afr J Physiother. 2019 Jun 3;75(1):904. doi: 10.4102/sajp.v75i1.904. eCollection 2019. PMID 31206094
- [Background] Lee H-J, Lee S-M. Effects of Schroth exercise therapy on curvature and body appearance of patients with lumbar idiopathic scoliosis. Physical Therapy Rehabilitation Science. 2020;9(4):230-7.
- [Background] Liu D, Yang Y, Yu X, Yang J, Xuan X, Yang J, Huang Z. Effects of Specific Exercise Therapy on Adolescent Patients With Idiopathic Scoliosis: A Prospective Controlled Cohort Study. Spine (Phila Pa 1976). 2020 Aug 1;45(15):1039-1046. doi: 10.1097/BRS.0000000000003451. PMID 32675606
- [Background] Kuru T, Yeldan I, Dereli EE, Ozdincler AR, Dikici F, Colak I. The efficacy of three-dimensional Schroth exercises in adolescent idiopathic scoliosis: a randomised controlled clinical trial. Clin Rehabil. 2016 Feb;30(2):181-90. doi: 10.1177/0269215515575745. Epub 2015 Mar 16. PMID 25780260
- [Background] Lee BK. Influence of the proprioceptive neuromuscular facilitation exercise programs on idiopathic scoliosis patient in the early 20s in terms of curves and balancing abilities: single case study. J Exerc Rehabil. 2016 Dec 31;12(6):567-574. doi: 10.12965/jer.1632796.398. eCollection 2016 Dec. PMID 28119879